CLINICAL TRIAL: NCT02414828
Title: A Phase II Double-Blind, Randomized, Placebo-controlled, Dose Escalation Study to Evaluate the Safety of AERAS-402 in Adults Recently Treated for Pulmonary Tuberculosis
Brief Title: A Study to Evaluate the Safety of AERAS-402 in Adults Recently Treated for Pulmonary TB
Acronym: C-010-402
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aeras (Other)
Collaborators: Crucell Holland BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C-010-402
Record Dates: First submitted 2015-04-08; First posted 2015-04-13 (Estimated); Results first posted 2016-05-04 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-04

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — AERAS-402

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): Placebo control: 1.0 mL sterile buffer containing 20 mM Tris buffer, 2 mM MgCl2, 25 mM NaCl, 10% w/v sucrose, 0.02% w/v PS-80 (polysorbate-80, non animal source) and water.
  Interventions: Biological: Placebo
- AERAS-402 3 x 10^8 vp (Experimental): AERAS-402: 1.0 mL containing 3 x 10^8 vp/mL suspended in 20 mM Tris buffer, 2 mM MgCl2, 25 mM NaCl, 10% w/v sucrose, 0.02% w/v PS-80 (polysorbate-80, non animal source) and water.
  Interventions: Biological: AERAS-402 3 x 10^8 vp
- AERAS-402 3 x 10^9 vp (Experimental): AERAS-402: 1.0 mL containing 3 x 10^9 vp/mL suspended in 20 mM Tris buffer, 2 mM MgCl2, 25 mM NaCl, 10% w/v sucrose, 0.02% w/v PS-80 (polysorbate-80, non animal source) and water.
  Interventions: Biological: AERAS-402 3 x 10^9 vp
- AERAS-402 3 x 10^10 vp (Experimental): AERAS-402: 1.0 mL containing 3 x 10^10 vp/mL suspended in 20 mM Tris buffer, 2 mM MgCl2, 25 mM NaCl, 10% w/v sucrose, 0.02% w/v PS-80 (polysorbate-80, non animal source) and water.
  Interventions: Biological: AERAS-402 3 x 10^10 vp

INTERVENTIONS:
Biological: Placebo — This is the identical buffer solution in which AERAS-402 is formulated. The placebo (1.0 mL volume) was administered by intramuscular (IM) injection to the deltoid area on Study Day 0 for groups 1 and 2 and Study Day 0 and 42 for group 3.
  Other Names: Sterile buffer
  Arms: Placebo
Biological: AERAS-402 3 x 10^8 vp — AERAS-402 was administered by single intramuscular (IM) injection to the deltoid area on Study Day 0
  Other Names: AERAS-402
  Arms: AERAS-402 3 x 10^8 vp
Biological: AERAS-402 3 x 10^9 vp — AERAS-402 was administered by single intramuscular (IM) injection to the deltoid area on Study Day 0
  Other Names: AERAS-402
  Arms: AERAS-402 3 x 10^9 vp
Biological: AERAS-402 3 x 10^10 vp — AERAS-402 was administered by intramuscular (IM) injection to the deltoid area on Study Days 0 and 42.
  Other Names: AERAS-402
  Arms: AERAS-402 3 x 10^10 vp

SUMMARY:
This was a double-blind, randomized, placebo-controlled dose-escalation study in adults recently treated for pulmonary TB. The dose of AERAS-402 increased in successive dose groups. Enrollment into a dose group was sequential. Enrollees were stratified based on time from the start of TB treatment. The "on-TB-treatment" stratum started TB treatment between 1 and 4 months (30 to 120 calendar days) prior to Study Day 0. The "post-TB-treatment" stratum started TB treatment at least 12 months (360 calendar days) prior to Study Day 0. Subjects were randomized to receive a placebo or AERAS-402 vaccine. In Dose Groups 1 and 2, subjects were randomized to receive a single injection of AERAS-402 or placebo. Dose Group 3 subjects were randomized to receive two injections on study day 0 and study day 42 of AERAS-402 or placebo.

DETAILED DESCRIPTION:
A total of 72 subjects were randomized into the study. Subjects were stratified, based on time from the start of TB treatment, into the 'on-TB-treatment' stratum (TB treatment started between 1 and 4 months prior to Study Day 0) or the 'post-TB-treatment' stratum (TB treatment started at least 12 months before Study Day 0). In the on-TB-treatment stratum, 36 subjects were randomized to receive AERAS-402 or placebo as follows: 1 or 2 doses of placebo (N=5); 1 dose of AERAS-402 at 3 x 10^8 vp (N=5) or 3 x 10^9 vp (N=10), or 2 doses of AERAS-402 at 3 x 10^10 vp (N=16). In the post-TB-treatment stratum, 36 subjects were randomized to receive AERAS-402 or placebo as follows: 1 or 2 doses of placebo (N=6); 1 dose of AERAS-402 at 3 x 10^8 vp (N=5) or 3 x 109 vp (N=10), or 2 doses of AERAS-402 at 3 x 10^10 vp (N=15).

ELIGIBILITY:
Inclusion Criteria:

1. Is male or female.
2. Is age 18 through 45 years on Study Day 0.
3. Has completed the written informed consent process.
4. Has a history of pulmonary tuberculosis diagnosed by either a sputum smear positive for acid-fast bacilli (AFB) or a sputum culture positive for Mtb.
5. Has initiated effective chemotherapy for tuberculosis between one month (30 days) and four months (120 days) before Study Day 0, with improvement in clinical signs and/or symptoms of disease,

   OR:

   has initiated effective chemotherapy for tuberculosis at least 12 months (360 days) before Study Day 0, and is considered cured.
6. For subjects currently receiving chemotherapy for tuberculosis they must have been fully compliant with previously prescribed tuberculosis therapy and agree to complete currently prescribed tuberculosis therapy.
7. Agrees to avoid elective surgery for the full duration of the study.
8. For female subjects: agrees to avoid pregnancy for the full duration of the study.
9. Agrees to stay in contact with the study site for the full duration of the study, providing updated contact information as necessary, and has no current plans to move from the study area during the duration of the study.
10. Has completed simultaneous enrollment in Aeras Vaccine Development Registry Protocol.

Exclusion Criteria:

1. Fever ≥37.5°C.
2. Evidence of a new acute illness that may compromise the safety of the subject in the study.
3. Evidence of any significant active infection other than tuberculosis.
4. Evidence of central nervous system tuberculosis or pleural tuberculosis.
5. Previous medical history that may compromise the safety of the subject in the study, including but not limited to: severe impairment of pulmonary function from tuberculosis infection or other pulmonary disease; chronic illness with signs of cardiac or renal failure; suspected progressive neurological disease; or uncontrolled epilepsy or infantile spasms.
6. Evidence of any systemic disease or any acute or chronic illness that may interfere with the evaluation of the safety of the vaccine.
7. History or laboratory evidence of any past, present or future possible immunodeficiency state, including but not limited to any laboratory indication of HIV-1 infection.
8. History of allergic disease or reactions likely to be exacerbated by any component of the study vaccine.
9. Received any investigational drug therapy or vaccine within 182 days before the first dose of study vaccine in this protocol.
10. Received any adenovirus-based vaccine previously.
11. For female subjects: Currently pregnant, lactating/nursing, or a positive serum or urine βhCG
12. Severe anemia, defined as a hemoglobin less than 10 g/dL or a hematocrit less than 30 percent.
13. Urine toxicology screen positive for opiates, cocaine, or amphetamines.
14. Anal intercourse with another man at least one time (with or without condoms).
15. Exchange of goods, money, services or drugs for sex.
16. Use of intravenous drugs.
17. Sexual intercourse or genital contact within the last 12 months with a known HIV positive individual.
18. Vaginal intercourse within the last 12 months without use of a condom with a known user of intravenous drugs.
19. Oral to genital contact within the last 12 months with a known user of intravenous drugs.
20. Vaginal intercourse within the last 12 months without use of a condom with an individual known to have more than one sex partner.
21. Oral to genital contact within the last 12 months with an individual known to have more than one sex partner.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2008-10; Primary Completion 2010-07 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Bateman, MD, Principal Investigator — University of Cape Town Lung Institute Pty (Ltd)
Locations (1):
- University of Cape Town Lung Institute Pty (Ltd), Cape Town, Mowbray, South Africa

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] van Zyl-Smit RN, Esmail A, Bateman ME, Dawson R, Goldin J, van Rikxoort E, Douoguih M, Pau MG, Sadoff JC, McClain JB, Snowden MA, Benko J, Hokey DA, Rutkowski KT, Graves A, Shepherd B, Ishmukhamedov S, Kagina BMN, Abel B, Hanekom WA, Scriba TJ, Bateman ED. Safety and Immunogenicity of Adenovirus 35 Tuberculosis Vaccine Candidate in Adults with Active or Previous Tuberculosis. A Randomized Trial. Am J Respir Crit Care Med. 2017 May 1;195(9):1171-1180. doi: 10.1164/rccm.201603-0654OC. PMID 28060545

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Sterile buffer, Intramuscular (IM)
- AERAS-402 3 x 10^8 vp; AERAS-402 3 x 10^9 vp: AERAS-402, 1 x IM, study day 0
- AERAS-402 3 x 10^10 vp: AERAS-402, 2 x IM, study days 0 and 42
Period: Overall Study
Arm/Group | Placebo | AERAS-402 3 x 10^8 vp | AERAS-402 3 x 10^9 vp | AERAS-402 3 x 10^10 vp
Started | 11 | 10 | 20 | 31
Completed | 11 | 9 | 19 | 29
Not Completed | 0 | 1 | 1 | 2
Not completed — Lost to Follow-up | 0 | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | AERAS-402 3 x 10^8 vp | AERAS-402 3 x 10^9 vp | AERAS-402 3 x 10^10 vp | Total
Number analyzed (Participants) | 11 | 10 | 20 | 31 | 72
Age, Customized [Number; unit: years]
  18-30 years | 6 | 5 | 11 | 20 | 42
  31-40 years | 4 | 2 | 5 | 9 | 20
  41-45 years | 1 | 3 | 4 | 2 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 14 | 16 | 41
  Male | 6 | 4 | 6 | 15 | 31
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 0 | 0 | 0 | 0 | 0
  Black | 1 | 3 | 9 | 9 | 22
  Coloured | 10 | 6 | 11 | 21 | 48
  White | 0 | 1 | 0 | 1 | 2
TB Treatment Status [Number; unit: participants] — "On TB Treatment" stratum started TB treatment between 1 and 4 months prior to Study Day 0. The "Post TB Treatment" stratum started TB treatment at least 12 months prior to Study Day 0
  participants
    On TB Treatment | 5 | 5 | 10 | 16 | 36
    Post TB Treatment | 6 | 5 | 10 | 15 | 36
History of Smoking [Number; unit: participants]
  Yes - History of smoking | 11 | 6 | 14 | 20 | 51
  No - History of Smoking | 0 | 4 | 6 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited and Unsolicited AEs
Description: All adverse events will be summarized to examine the relationship between dose levels including number (percentage) of solicited and unsolicited adverse events (AEs), and number (percentage) of subjects with newly abnormal post-vaccination laboratory values based on predefined toxicity criteria.
Time Frame: 182 days
Measure: Number; unit: participants
Arm/Group | Placebo | AERAS-402 3 x 10^8 vp | AERAS-402 3 x 10^9 vp | AERAS-402 3 x 10^10 vp
Number analyzed (Participants) | 11 | 10 | 20 | 31
participants | 11 | 10 | 20 | 30

2. Secondary Outcome: Immunogenicity of AERAS-402 Based on the Percentage of CD4 Cells of Participants in the "on TB Treatment" Stratum
Description: Assessment of immune response to AERAS-402 was based on the percentage of CD4 and CD8 T cells producing any combination of three cytokines (IFN-γ, TNF-α, and/or IL-2) following stimulation with mycobacterial peptide pools derived from and representing the entire amino acid sequences of mycobacterial antigens Ag85A, Ag85B, and TB10.4. Responses were measured by the intracellular cytokine staining (ICS) assay using flow cytometry.
Time Frame: 42 days post dose
Measure: Median (95% Confidence Interval); unit: percentage of T Cell response
Groups:
- Placebo: Sterile buffer, IM
Arm/Group | Placebo | AERAS-402 3 x 10^8 vp | AERAS-402 3 x 10^9 vp | AERAS-402 3 x 10^10 vp
Number analyzed (Participants) | 5 | 5 | 10 | 16
percentage of T Cell response
  On TB Treatment CD4 Ag85A Day 0 | 0.025 [0.025 to 0.168] | 0.025 [0.025 to 0.025] | 0.025 [0.025 to 0.062] | 0.025 [0.025 to 0.025]
  On TB Treatment CD4 Ag85A Day 42 | 0.025 [0.025 to 0.025] | 0.056 [0.025 to 0.112] | 0.057 [0.025 to 0.176] | 0.061 [0.025 to 0.121]
  On TB Treatment CD4 Ag85A Day 84 | 0.025 [0.025 to 0.025] | NA [NA to NA] — No second dose given | NA [NA to NA] — No second dose given | 0.072 [0.025 to 0.228]
  On TB Treatment CD4 Ag85B Day 0 | 0.025 [0.025 to 0.097] | 0.025 [0.025 to 0.025] | 0.025 [0.025 to 0.085] | 0.025 [0.025 to 0.093]
  On TB Treatment CD4 Ag85B Day 42 | 0.025 [0.025 to 0.025] | 0.025 [0.025 to 0.112] | 0.052 [0.025 to 0.175] | 0.082 [0.025 to 0.160]
  On TB Treatment CD4 Ag85B Day 84 | 0.233 [0.164 to 0.303] | NA [NA to NA] — No second dose given | NA [NA to NA] — No second dose given | 0.489 [0.153 to 0.789]
  On TB Treatment CD4 TB10.4 Day 0 | 0.068 [0.025 to 0.143] | 0.025 [0.025 to 0.025] | 0.063 [0.025 to 0.115] | 0.025 [0.025 to 0.025]
  On TB Treatment CD4 TB10.4 Day 42 | 0.025 [0.025 to 0.025] | 0.025 [0.025 to 0.223] | 0.053 [0.025 to 0.064] | 0.025 [0.025 to 0.084]
  On TB Treatment CD4 TB10.4 Day 84 | 0.120 [0.025 to 0.216] | NA [NA to NA] — No second dose given | NA [NA to NA] — No second dose given | 0.043 [0.025 to 0.094]

3. Primary Outcome: Forced Expiratory Volume in One Second (FEV1)
Description: Maximum number of subjects with deterioration >10% from baseline, at any time point. in forced expiratory volume in one second (FEV1)
Time Frame: 182 days
Population: Subjects who were evaluated.
Measure: Number; unit: participants
Arm/Group | Placebo | AERAS-402 3 x 10^8 vp | AERAS-402 3 x 10^9 vp | AERAS-402 3 x 10^10 vp
Number analyzed (Participants) | 5 | 10 | 20 | 29
participants
  On TB Treatment | 1 | 2 | 0 | 3
  Post TB Treatment | 1 | 3 | 1 | 5

4. Primary Outcome: Forced Vital Capacity (FVC)
Description: Maximum number of subjects with deterioration >10% from baseline, at any time point, in forced vital capacity (FVC)
Time Frame: 182 days
Population: Subjects who were evaluated.
Measure: Number; unit: participants
Arm/Group | Placebo | AERAS-402 3 x 10^8 vp | AERAS-402 3 x 10^9 vp | AERAS-402 3 x 10^10 vp
Number analyzed (Participants) | 5 | 10 | 20 | 29
participants
  On TB Treatment | 1 | 2 | 0 | 1
  Post TB Treatment | 1 | 3 | 3 | 4

5. Primary Outcome: Diffusing Capacity of the Lung for Carbon Monoxide (DLCO)
Description: Maximum number of subjects with deterioration >15% from baseline, at any time point, in diffusing capacity of the lung for carbon monoxide (DLCO)
Time Frame: 182 Days
Population: Subjects who were evaluated.
Measure: Number; unit: participants
Arm/Group | Placebo | AERAS-402 3 x 10^8 vp | AERAS-402 3 x 10^9 vp | AERAS-402 3 x 10^10 vp
Number analyzed (Participants) | 5 | 9 | 20 | 30
participants
  On TB Treatment | 1 | 3 | 0 | 5
  Post TB Treatment | 1 | 2 | 2 | 7

6. Secondary Outcome: Immunogenicity of AERAS-402 Based on the Percentage of CD8 Cells of Participants in the "on TB Treatment" Stratum
Description: as for outcome 2
Time Frame: 42 days post dose
Measure: Median (95% Confidence Interval); unit: percentage of T Cell response
Arm/Group | Placebo | AERAS-402 3 x 10^8 vp | AERAS-402 3 x 10^9 vp | AERAS-402 3 x 10^10 vp
Number analyzed (Participants) | 5 | 5 | 10 | 16
percentage of T Cell response
  On TB Treatment CD8 Ag85A Day 0 | 0.025 [0.025 to 0.025] | 0.025 [0.025 to 0.025] | 0.025 [0.025 to 0.025] | 0.025 [0.025 to 0.210]
  On TB Treatment CD8 Ag85A Day 42 | 0.025 [0.025 to 0.070] | 0.085 [0.025 to 0.258] | 0.301 [0.081 to 2.049] | 0.076 [0.025 to 0.584]
  On TB Treatment CD8 Ag85A Day 84 | 0.025 [0.025 to 0.025] | NA [NA to NA] — No second dose given | NA [NA to NA] — No second dose given | 0.169 [0.025 to 2.340]
  On TB Treatment CD8 Ag85B Day 0 | 0.025 [0.025 to 0.066] | 0.025 [0.025 to 0.025] | 0.025 [0.025 to 0.025] | 0.025 [0.025 to 0.481]
  On TB Treatment CD8 Ag85B Day 42 | 0.025 [0.025 to 0.083] | 0.089 [0.025 to 0.223] | 0.310 [0.104 to 2.352] | 0.125 [0.058 to 0.332]
  On TB Treatment CD8 Ag85B Day 84 | 0.080 [0.025 to 0.135] | NA [NA to NA] — No second dose given | NA [NA to NA] — No second dose given | 0.571 [0.364 to 2.239]
  On TB Treatment CD8 TB10.4 Day 0 | 0.025 [0.025 to 0.025] | 0.025 [0.025 to 0.025] | 0.025 [0.025 to 0.025] | 0.025 [0.025 to 0.142]
  On TB Treatment CD8 TB10.4 Day 42 | 0.025 [0.025 to 0.025] | 0.068 [0.025 to 0.078] | 0.025 [0.025 to 0.533] | 0.223 [0.025 to 0.505]
  On TB Treatment CD8 TB10.4 Day 84 | 0.025 [0.025 to 0.025] | NA [NA to NA] — No second dose given | NA [NA to NA] — No second dose given | 0.079 [0.025 to 0.315]

7. Secondary Outcome: Immunogenicity of AERAS-402 Based on the Percentage of CD4 Cells of Participants in the "Post TB Treatment" Stratum
Description: as for outcome 2
Time Frame: 42 days post dose
Measure: Median (95% Confidence Interval); unit: percentage of T Cell response
Arm/Group | Placebo | AERAS-402 3 x 10^8 vp | AERAS-402 3 x 10^9 vp | AERAS-402 3 x 10^10 vp
Number analyzed (Participants) | 6 | 5 | 10 | 15
percentage of T Cell response
  Post TB Treatment CD4 Ag85A Day 0 | 0.025 [0.025 to 0.025] | 0.025 [0.025 to 0.067] | 0.025 [0.025 to 0.060] | 0.025 [0.025 to 0.025]
  Post TB Treatment CD4 Ag85A Day 42 | 0.025 [0.025 to 0.025] | 0.056 [0.025 to 0.092] | 0.089 [0.025 to 0.148] | 0.057 [0.025 to 0.130]
  Post TB Treatment CD4 Ag85A Day 84 | 0.025 [0.025 to 0.025] | NA [NA to NA] — No second dose given | NA [NA to NA] — No second dose given | 0.091 [0.068 to 0.127]
  Post TB Treatment CD4 Ag85B Day 0 | 0.025 [0.025 to 0.290] | 0.025 [0.025 to 0.057] | 0.025 [0.025 to 0.064] | 0.025 [0.025 to 0.059]
  Post TB Treatment CD4 Ag85B Day 42 | 0.025 [0.025 to 0.237] | 0.038 [0.025 to 0.063] | 0.076 [0.025 to 0.146] | 0.105 [0.025 to 0.140]
  Post TB Treatment CD4 Ag85B Day 84 | 0.487 [0.025 to 0.657] | NA [NA to NA] — No second dose given | NA [NA to NA] — No second dose given | 0.547 [0.360 to 0.849]
  Post TB Treatment CD4 TB10.4 Day 0 | 0.025 [0.025 to 0.175] | 0.025 [0.025 to 0.093] | 0.040 [0.025 to 0.074] | 0.025 [0.025 to 0.068]
  Post TB Treatment CD4 TB10.4 Day 42 | 0.025 [0.025 to 0.163] | 0.025 [0.025 to 0.025] | 0.089 [0.025 to 0.174] | 0.025 [0.025 to 0.099]
  Post TB Treatment CD4 TB10.4 Day 84 | 0.025 [0.025 to 0.069] | NA [NA to NA] — No second dose given | NA [NA to NA] — No second dose given | 0.025 [0.025 to 0.103]

8. Secondary Outcome: Immunogenicity of AERAS-402 Based on the Percentage of CD8 Cells of Participants in the "Post TB Treatment" Stratum
Description: as for outcome 2
Time Frame: 42 days post dose
Measure: Median (95% Confidence Interval); unit: percentage of T Cell response
Arm/Group | Placebo | AERAS-402 3 x 10^8 vp | AERAS-402 3 x 10^9 vp | AERAS-402 3 x 10^10 vp
Number analyzed (Participants) | 6 | 5 | 10 | 15
percentage of T Cell response
  Post TB Treatment CD8 Ag85A Day 0 | 0.025 [0.025 to 0.025] | 0.025 [0.025 to 0.025] | 0.025 [0.025 to 0.057] | 0.025 [0.025 to 0.025]
  Post TB Treatment CD8 Ag85A Day 42 | 0.025 [0.025 to 0.025] | 0.584 [0.025 to 2.205] | 0.083 [0.025 to 2.037] | 0.054 [0.025 to 0.279]
  Post TB Treatment CD8 Ag85A Day 84 | 0.025 [0.025 to 0.025] | NA [NA to NA] — No second dose given | NA [NA to NA] — No second dose given | 0.400 [0.125 to 0.710]
  Post TB Treatment CD8 Ag85B Day 0 | 0.025 [0.025 to 0.228] | 0.025 [0.025 to 0.025] | 0.025 [0.025 to 0.025] | 0.025 [0.025 to 0.025]
  Post TB Treatment CD8 Ag85B Day 42 | 0.025 [0.025 to 0.193] | 0.439 [0.025 to 1.830] | 0.206 [0.025 to 1.945] | 0.169 [0.025 to 0.475]
  Post TB Treatment CD8 Ag85B Day 84 | 0.109 [0.025 to 0.393] | NA [NA to NA] — No second dose given | NA [NA to NA] — No second dose given | 0.673 [0.338 to 1.206]
  Post TB Treatment CD8 TB10.4 Day 0 | 0.025 [0.025 to 0.161] | 0.025 [0.025 to 0.025] | 0.025 [0.025 to 0.025] | 0.025 [0.025 to 0.025]
  Post TB Treatment CD8 TB10.4 Day 42 | 0.025 [0.025 to 0.094] | 0.025 [0.025 to 0.417] | 0.025 [0.025 to 0.285] | 0.025 [0.025 to 0.074]
  Post TB Treatment CD8 TB10.4 Day 84 | 0.025 [0.025 to 0.025] | NA [NA to NA] — No second dose given | NA [NA to NA] — No second dose given | 0.104 [0.025 to 0.251]

ADVERSE EVENTS:
Arm/Group | Placebo | AERAS-402 3 x 10^8 vp | AERAS-402 3 x 10^9 vp | AERAS-402 3 x 10^10 vp
Serious Adverse Events (participants affected / at risk) | 0/11 | 1/10 | 0/20 | 1/31
Other Adverse Events (participants affected / at risk) | 11/11 | 10/10 | 20/20 | 30/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=11) | AERAS-402 3 x 10^8 vp (N=10) | AERAS-402 3 x 10^9 vp (N=20) | AERAS-402 3 x 10^10 vp (N=31)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchioloalveolar carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=11) | AERAS-402 3 x 10^8 vp (N=10) | AERAS-402 3 x 10^9 vp (N=20) | AERAS-402 3 x 10^10 vp (N=31)
Bacteriuria (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 4 (6) | 2 (2) | 6 (6) | 6 (6)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Microcytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Polydipsia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight gain poor (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 2 (3) | 0 (0) | 0 (0) | 9 (10)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Labile blood pressure (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 1 (1) | 5 (5)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 0 (0) | 4 (4)
Rales (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 5 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 4 (4)
Bladder pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 3 (4) | 0 (0) | 2 (3) | 5 (7)
Fatigue (General disorders) | 2 (2) | 0 (0) | 1 (1) | 5 (6)
Injection site discharge (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 5 (5) | 1 (1) | 7 (7) | 15 (18)
Injection site haematoma (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 1 (1) | 1 (1) | 7 (8) | 20 (32)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 4 (4) | 5 (6)
Malaise (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Vessel puncture site haematoma (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 2 (2) | 2 (2) | 3 (3)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Blood pressure diastolic increased (Investigations) | 2 (2) | 1 (2) | 3 (5) | 2 (2)
Blood pressure systolic decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood pressure systolic increased (Investigations) | 2 (2) | 3 (3) | 1 (1) | 3 (3)
Blood urine present (Investigations) | 2 (2) | 0 (0) | 0 (0) | 9 (11)
Carbon monoxide diffusing capacity decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 14 (15)
Crystal urine present (Investigations) | 1 (2) | 0 (0) | 1 (1) | 2 (2)
False positive tuberculosis test (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Forced expiratory volume decreased (Investigations) | 2 (3) | 0 (0) | 0 (0) | 6 (9)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 6 (6)
Glucose urine (Investigations) | 1 (1) | 0 (0) | 3 (3) | 3 (3)
Haemoglobin decreased (Investigations) | 2 (2) | 3 (3) | 4 (4) | 9 (12)
Heart rate decreased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Heart rate increased (Investigations) | 4 (5) | 1 (1) | 1 (1) | 6 (8)
Lymphocyte count decreased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 4 (4)
Neutrophil count decreased (Investigations) | 2 (2) | 1 (2) | 3 (4) | 6 (7)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Protein urine (Investigations) | 6 (6) | 4 (4) | 6 (6) | 14 (20)
Red blood cell hypochromic morphology present (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Red blood cell morphology abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Red blood cells urine (Investigations) | 3 (3) | 0 (0) | 4 (4) | 10 (15)
Urine leukocyte esterase positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 8 (9)
Vital capacity decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
White blood cell count increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
White blood cells urine positive (Investigations) | 1 (1) | 0 (0) | 1 (1) | 6 (9)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Physical assault (Social circumstances) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No